CLINICAL TRIAL: NCT00547703
Title: Effect of Nortriptyline on Abdominal Pain/Discomfort and Quality of Life in Patients With Nonulcer Dyspepsia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants - only 5 since the study started
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Fernando Castro, Principal investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 8918
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Results first posted 2012-07-10 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Non Ulcer Dyspepsia
Keywords: Nonulcer dyspepsia; Functional dyspepsia; Antidepressant use in dyspepsia; Nortriptyline; Tricyclic antidepressants
MeSH Terms: interventions — Nortriptyline; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nortriptyline (Active Comparator): Patients in this group will receive Nortriptyline 25mg at night for 8 weeks.
  Interventions: Drug: Nortriptyline
- Sugar pill (Placebo Comparator): Patients in this group will receive an identical placebo capsule at night for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nortriptyline — Nortriptyline 25mg capsule, orally administered, every night for 8 weeks
  Other Names: Pamelor
  Arms: Nortriptyline
Drug: Placebo — An identical placebo capsule containing lactose, administered orally, every night for 8 weeks
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine if use of Nortriptyline will improve symptoms and quality of life in patients who have nonulcer dyspepsia.

DETAILED DESCRIPTION:
Nonulcer dyspepsia is a common complaint in clinical practice and its management should be based on the best evidence. Many clinical trials of nonulcer dyspepsia suffer from important weaknesses in trial design. This makes it difficult to determine whether truly efficacious therapies exist for this disorder.

Once a diagnosis of nonulcer dyspepsia is confirmed by normal endoscopy, a trial of therapy is commonly prescribed. However, the benefits of all therapies in this condition have been questioned. Small studies have suggested benefit in use of antidepressants such as Nortriptyline and even though the data is insufficient, antidepressants such as Nortriptyline are widely used in clinical practice largely due to lack of proven, reliable therapies for nonulcer dyspepsia.

Our hypothesis is that Nortriptyline will improve symptoms of nonulcer dyspepsia and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women
* Ages 18-65
* Meet Rome III criteria for functional dyspepsia
* Endoscopy within 1 year

Exclusion Criteria:

* Allergic reaction or history of adverse events with Nortriptyline or tricyclic antidepressants
* Organic cause found on physical examination
* Organic cause found on lab work: Complete Blood Count, Comprehensive Metabolic Panel, Thyroid stimulating hormone, Tissue transglutaminase Immunoglobulin A
* Predominantly Gastroesophageal reflux symptoms
* Current Helicobacter pylori infection
* History of Peptic ulcer disease
* Non steroidal antiinflammatory use use > 2x/wk
* Pregnant or planning pregnancy
* History of major depression
* Abdominal surgery in the last year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-02; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Castro, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mertz H, Fass R, Kodner A, Yan-Go F, Fullerton S, Mayer EA. Effect of amitriptyline on symptoms, sleep, and visceral perception in patients with functional dyspepsia. Am J Gastroenterol. 1998 Feb;93(2):160-5. doi: 10.1111/j.1572-0241.1998.00160.x. PMID 9468233
- [Background] Tanum L, Malt UF. A new pharmacologic treatment of functional gastrointestinal disorder. A double-blind placebo-controlled study with mianserin. Scand J Gastroenterol. 1996 Apr;31(4):318-25. doi: 10.3109/00365529609006404. PMID 8726297
- [Background] Wiklund IK, Junghard O, Grace E, Talley NJ, Kamm M, Veldhuyzen van Zanten S, Pare P, Chiba N, Leddin DS, Bigard MA, Colin R, Schoenfeld P. Quality of Life in Reflux and Dyspepsia patients. Psychometric documentation of a new disease-specific questionnaire (QOLRAD). Eur J Surg Suppl. 1998;(583):41-9. PMID 10027672
- [Background] Veldhuyzen van Zanten SJ, Chiba N, Armstrong D, Barkun AN, Thomson AB, Mann V, Escobedo S, Chakraborty B, Nevin K. Validation of a 7-point Global Overall Symptom scale to measure the severity of dyspepsia symptoms in clinical trials. Aliment Pharmacol Ther. 2006 Feb 15;23(4):521-9. doi: 10.1111/j.1365-2036.2006.02774.x. PMID 16441473
- [Background] Hojo M, Miwa H, Yokoyama T, Ohkusa T, Nagahara A, Kawabe M, Asaoka D, Izumi Y, Sato N. Treatment of functional dyspepsia with antianxiety or antidepressive agents: systematic review. J Gastroenterol. 2005 Nov;40(11):1036-42. doi: 10.1007/s00535-005-1687-8. PMID 16322947
- [Background] Veldhuyzen van Zanten SJ, Cleary C, Talley NJ, Peterson TC, Nyren O, Bradley LA, Verlinden M, Tytgat GN. Drug treatment of functional dyspepsia: a systematic analysis of trial methodology with recommendations for design of future trials. Am J Gastroenterol. 1996 Apr;91(4):660-73. PMID 8677926
- [Background] Talley NJ, Vakil N; Practice Parameters Committee of the American College of Gastroenterology. Guidelines for the management of dyspepsia. Am J Gastroenterol. 2005 Oct;100(10):2324-37. doi: 10.1111/j.1572-0241.2005.00225.x. PMID 16181387
- [Background] Jackson JL, O'Malley PG, Tomkins G, Balden E, Santoro J, Kroenke K. Treatment of functional gastrointestinal disorders with antidepressant medications: a meta-analysis. Am J Med. 2000 Jan;108(1):65-72. doi: 10.1016/s0002-9343(99)00299-5. PMID 11059442
- [Background] Talley NJ. Therapeutic options in nonulcer dyspepsia. J Clin Gastroenterol. 2001 Apr;32(4):286-93. doi: 10.1097/00004836-200104000-00004. PMID 11276271
- [Background] Talley NJ, Fullerton S, Junghard O, Wiklund I. Quality of life in patients with endoscopy-negative heartburn: reliability and sensitivity of disease-specific instruments. Am J Gastroenterol. 2001 Jul;96(7):1998-2004. doi: 10.1111/j.1572-0241.2001.03932.x. PMID 11467624
- [Background] Design of Treatment Trials Committee; Irvine EJ, Whitehead WE, Chey WD, Matsueda K, Shaw M, Talley NJ, Veldhuyzen van Zanten SJ. Design of treatment trials for functional gastrointestinal disorders. Gastroenterology. 2006 Apr;130(5):1538-51. doi: 10.1053/j.gastro.2005.11.058. PMID 16678567
- [Background] Veldhuyzen van Zanten SJ, Talley NJ, Bytzer P, Klein KB, Whorwell PJ, Zinsmeister AR. Design of treatment trials for functional gastrointestinal disorders. Gut. 1999 Sep;45 Suppl 2(Suppl 2):II69-77. doi: 10.1136/gut.45.2008.ii69. PMID 10457048
- [Background] Moayyedi P, Delaney BC, Vakil N, Forman D, Talley NJ. The efficacy of proton pump inhibitors in nonulcer dyspepsia: a systematic review and economic analysis. Gastroenterology. 2004 Nov;127(5):1329-37. doi: 10.1053/j.gastro.2004.08.026. PMID 15521002

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients in this group will receive an identical placebo capsule at night for 8 weeks.
Period: Overall Study
Arm/Group | Nortriptyline | Placebo
Started | 4 | 1
Completed | 3 | 1
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nortriptyline | Placebo | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (4) | 43 (0) | 42 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Question on Whether Patient Has Had Adequate Relief of Abdominal Pain or Discomfort Reported by a Simple Yes or no Answer.
Description: Patient would answer yes or no to a simple question asking whether they had adequate relief of abdominal pain or discomfort. This was measured at weeks 2,4 and 8 of the study but only week 8 was reported. What is being reported is the number of participants who answered yes.
Time Frame: 8 weeks
Population: All patients who completed the 8 weeks of the study
Measure: Number; unit: participants
Arm/Group | Nortriptyline | Placebo
Number analyzed (Participants) | 3 | 1
participants | 2 | 1

2. Secondary Outcome: QOLRAD Questionaire for Patients With Upper Abdominal Symptoms
Description: Patients were administered the validated QOLRAD questionnaire on quality of life to assess if nortriptyline improves quality of life in patients with nonulcer dyspepsia
Time Frame: 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Side Effects
Description: To assess frequency of side effects in patients receiving Nortriptyline for nonulcer dyspepsia. Patients were asked about side effects on each office visit and ask to call for significant side effects.
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Nortriptyline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 2/3 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nortriptyline (N=3) | Placebo (N=1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
We were unable to recruit an adequate number of patients to make any meaningful conclusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes